CLINICAL TRIAL: NCT02461953
Title: HA130 Hemoperfusion Apparatus Combined Hemodialysis to Improve Quality of Life in Patients Undergoing Maintenance Hemodialysis：A Perspective, Randomized, Controlled Multicenter Clinical Study
Brief Title: Combination of Hemodialysis With Hemoperfusion：A Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiangmei Chen, Professor,Chief physician,Academician of Chinese Academy of Engineering,Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-011
Record Dates: First submitted 2015-06-02; First posted 2015-06-03 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Renal Dialysis; Hemoperfusion; Quality of Life
Keywords: hemodialysis; hemoperfusion; quality of life

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- low flux hemodialysis (Experimental): low flux hemodialysis alone, 3 times a week, 4 hours per session
  Interventions: Device: low flux dialyzer
- high flux hemodialysis (Experimental): high flux hemodialysis alone, 3 times a week, 4 hours per session
  Interventions: Device: high flux dialyzer
- low flux hemodialysis + hemoperfusion (Experimental): low flux hemodialysis 2times a week and the HD+HP once a week
  Interventions: Device: hemoperfusion apparatus; Device: low flux dialyzer
- high flux hemodialysis + hemoperfusion (Experimental): high flux hemodialysis 2times a week and the HD+HP once a week
  Interventions: Device: hemoperfusion apparatus; Device: high flux dialyzer

INTERVENTIONS:
Device: hemoperfusion apparatus
  Other Names: hemoperfusion apparatus(HA-130;Jafron Biomedical Co., Ltd）
  Arms: high flux hemodialysis + hemoperfusion; low flux hemodialysis + hemoperfusion
Device: low flux dialyzer
  Arms: low flux hemodialysis; low flux hemodialysis + hemoperfusion
Device: high flux dialyzer
  Arms: high flux hemodialysis; high flux hemodialysis + hemoperfusion

SUMMARY:
This study is a prospective, randomized, controlled multicenter clinical study. The aim of the study is to investigate whether the combination of maintenance hemodialysis (MHD) with hemoperfusion (HP) could improve the clearance rate of middle and large molecule uremic toxins so as to improve the quality of life of MHD patients and reduce their mortality rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18, male or female
2. Maintenance hemodialysis duration>3 months
3. Regular hemodialysis,3 times a week,4 hours per session
4. Vascular access unlimited
5. iPTH≥300pg/ml
6. Sign the written informed consent

Exclusion Criteria:

1. Allergic to dialysis equipment
2. PLT<60×10^9/L
3. Blood flow<200ml/min
4. Serum albumin<30g/L
5. Kt/V<1.2
6. iPTH>800pg/ml
7. Hemodiafiltration
8. Coagulation disorder, severe bleeding tendency, with active bleeding
9. Severe hypotension, severe cardiopulmonary insufficiency
10. Under other drug trial
11. Acute infection, severe heart, lung, liver, nervous diseases, malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Clearance rate of uremic toxins | 0,3,6,12 months

SECONDARY OUTCOMES:
Evaluation of quality of life | 0,3,6,12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China